CLINICAL TRIAL: NCT06226766
Title: Phase I/II Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of JSKN033 in Patients With Advanced or Metastatic Solid Malignant Tumors
Brief Title: JSKN033 in Patients With Advanced or Metastatic Solid Malignant Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the decision is based on a strategic realignment of our clinical trial priorities to optimize the overall development pathway for JSKN033
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JSKN033-101
Record Dates: First submitted 2023-12-22; First posted 2024-01-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose escalation/expansion (Experimental): The dose escalation phase will utilize single patient accelerated dose titration (ADT) for dose level 1 (1.1 mg/kg , SC, QW) and dose level 2 (2.3 mg/kg, SC, QW), followed by dose level 3 (4.5 mg/kg, SC, QW), dose level 4 (5.6 mg/kg, SC, QW) and dose level 5 (6.7 mg/kg, SC,QW), which will all be enrolled and monitored using the "3+3" design, aimed at determining the MTD/RP2D of JSKN033.
  After or during dose escalation, SMC will select 1-2 dose levels to expand with 10-30 additional patients with gastrointestinal tumor with HER2 expression each dose level for further exploration of the efficacy and safety of JSKN033.
  Interventions: Drug: JSKN033 Injection

INTERVENTIONS:
Drug: JSKN033 Injection — JSKN033 is a combination drug product comprised of JSKN003 and envafolimab for subcutaneous injection.

SUMMARY:
This study is an open-label, multicenter, first-in-human, Phase I/II (dose escalation and dose expansion) study to evaluate the safety, tolerability, PK, immunogenicity and efficacy of JSKN033 in patients with advanced unresectable or metastatic solid malignant tumors that are expected to be HER2 expression (IHC ≥ 1+).

DETAILED DESCRIPTION:
This study is an open label, multicenter, first in human, Phase I/II (dose escalation and dose expansion) study to evaluate the safety, tolerability, PK, immunogenicity and efficacy of JSKN033 in patients with advanced unresectable or metastatic solid malignant tumors that are expected to be HER2 expression.

JSKN033 is a combination drug product comprised of JSKN003 and envafolimab for subcutaneous injection.

Phase I will be a dose escalation phase - Participants will be enrolled to receive 1.1 mg/kg , 2.3 mg/kg, 4.5 mg/kg, 5.6 mg/kg or 6.7 mg/kg, once a week.

Phase II will be a dose expansion phase - After/during dose escalation, SMC will select 1-2 dose levels to expand with additional patients with gastrointestinal tumor with HER2 expression each dose level for further exploration of the efficacy and safety of JSKN033. Once treatment is discontinued, participants will be followed up every 12 weeks for any AEs and alternative anti-cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent form (ICF) for the trial.
2. Male or female, 18 years of age or older; willing and able to complete all required procedures of study.
3. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1, and life expectancy ≥ 12 weeks.
4. Must have a pathologically documented advanced unresectable or metastatic solid malignant tumor (gastrointestinal tumor for dose expansion phase) with HER2 expression (IHC ≥1+) that is refractory to or intolerable with standard treatment, or for which no effective standard treatment is available. HER2 mutation in patients with NSCLC is also regarded as HER2 expression.
5. Baseline measurable disease according to RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
6. Adequate organ function assessed within 7 days prior to first trial treatment [had not received blood transfusion, erythropoietin (EPO), granulocyte colony stimulating factor (G-CSF) or other relevant medical support within 14 days before the administration of the investigational product].
7. Have adequate treatment washout period before first dose.
8. Have LVEF ≥50% by either echo cardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days prior to first dose.
9. Female or male patients of childbearing potential should be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 180 days after completion of study treatment. Female of childbearing potential should have a negative pregnancy test within 7 days prior to first trial treatment (childbearing potential is defined as premenopausal females without documented tubal ligation or hysterectomy, or postmenopausal females within 1 year).

Exclusion Criteria:

1. Patients with untreated active brain metastases or meningeal or spinal cord metastases are excluded. If the subject has received treatment for brain metastases and the metastases are stable (as evidenced by brain imaging within 28 days prior to study treatment showing stable disease, no new lesions, and no new neurological symptoms, and no requirement for steroids for at least 14 days prior to study treatment), they may be eligible for enrollment.
2. Concurrent malignancy within 5 years prior to first dose other than adequately treated cervical carcinoma-in-situ, localized squamous cell cancer of the skin, basal cell carcinoma, prostate cancer, thyroid cancer not requiring treatment, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
3. Prior treatment with an antibody-drug conjugate (ADC) which consists of a topoisomerase I inhibitor derivative.
4. History of uncontrolled concurrent illness.
5. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids or current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by image at screening.
6. Previous severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) infection either suspected or confirmed within 4 weeks prior to screening. Acute symptoms will be excluded, or must have resolved and based on investigator assessment, there are no sequela that would place participant at a higher risk of receiving investigational treatment.
7. Patients with ascites, pleural effusion, pericardial effusion which cannot be controlled by appropriate interventions.
8. Have unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia, grade 2 hypoparathyroidism) related to prior anticancer therapy and stable anemia not yet resolved to grade ≤ 1 (NCI-CTCAEV5.0).
9. Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. A brief course of corticosteroids for the prophylaxis (e.g., contrast dye allergy) or treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.
10. History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or excipients in JSKN033 drug formulation.
11. Prior history of anti-HER2 therapy induced angioedema, or severe hypotension and Severe allergic reactions to other antibody drugs or topoisomerase I inhibitors.
12. Other conditions that, in the investigators' opinion, would make patients inappropriate to participate in this study, such as a history of mental illness, alcoholism or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), serious adverse events (SAEs), assessed by CTCAE V5.0 | Postdose of last participant up to 1 year
  Clinically significant changes in physical examination findings, vital sign measurements, standard clinical laboratory parameters, 12-lead electrocardiogram (ECG) parameters, ECHO cardiography or multiple-gated acquisition (MUGA) scan findings will be recorded as AEs.
RP2D( recommend Phase II dose) | Postdose of last participant up to 1 year
  To determine RP2D of JSKN033
DLTs （Dose-limiting toxicities） | Baseline up to 21 days after the first dose
  DLTs are defined as side effects of a drug or other treatment that are serious enough to prevent an increase in dose or level of that treatment.
Objective Response Rate (ORR) Following Treatment With JSKN033 in Participants With Advanced Solid Malignant Tumors | From 6 weeks postdose of last participant up to 1 years
  Objective response rate (ORR) by investigators' review was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Postdose of last participant up to 1 year
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab
Time at which Cmax is reached (Tmax) | Postdose of last participant up to 1 year
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab
Area under the drug concentration-time curve (AUC) to the last observable concentration (AUClast) | Postdose of last participant up to 1 year
  Categories: JSKN003, total antibody (Tab) , payload of JSKN003 and envafolimab
Progression-Free Survival (PFS) Following Treatment With JSKN033 in Participants | Postdose of last participant up to 1 year
  PFS by investigator assessment is defined as the time from first dose of study drug to disease progression(as per RECIST v1.1) or death
Duration of Response (DoR) Following Treatment With JSKN033 in Participants | Postdose of last participant up to 1 year
  DOR is defined as the time from assessment of complete response or partial response to disease progression or death in patients who achieve complete or partial response.
Overall Survival (OS) Following Treatment With JSKN033 in Participants | Postdose of last participant up to 1 year
  OS is defined as the time from first dose of study drug to death due to any cause. If there is no death reported for a subject before the data cutoff for OS analysis, OS will be censored at the last contact date at which the subject is known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, Principal Investigator — Scientia Clinical Research
Locations (1):
- Scientia Clinical Research, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No